CLINICAL TRIAL: NCT02802397
Title: AROPE : Early Ovarian Reserve Decreased : Impact of Exposure to Persistent Endocrine Disruptors and Organic Solvents
Acronym: AROPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC16_9748_AROPE; 2016-A00307-44 (Registry Identifier: ANSM); 16/14-1012 (Other: CPP Ouest V (Rennes)); 160295B-22 (Other: ANSM)
Record Dates: First submitted 2016-05-17; First posted 2016-06-16 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Female Infertility
Keywords: Early ovarian reserve decreased
MeSH Terms: conditions — Infertility, Female | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cases (Other): Cases and controls will benefit, as usual in France concerning infertility etiology examinations, of a follicle antral count by transvaginal ultrasound and AMH measurement.
  At baseline, physicians will complete a short questionnaire to check the inclusion criterion, the results of the measurement of follicle count and hormone measurement (including AMH). Cases and controls will respond to self-administered questionnaire at inclusion with information about their medical history, their demographics, their tobacco and alcohol consumption, their occupation and products handled in the workplace. Blood samples (for measure of persistent organic pollutants and heavy metals) and urine (for measure of metabolites of glycol ethers) will be collect at baseline. Occupational exposures to solvents will be defined using job exposures matrices. The risk of decreased ovarian reserve will be analyzed using logistic regressions for each exposure of interest adjusting for potential confounders.
  Interventions: Other: Self-administered questionnaire and blood and urine samples
- Controls (Other): Cases and controls will benefit, as usual in France concerning infertility etiology examinations, of a follicle antral count by transvaginal ultrasound and AMH measurement.
  At baseline, physicians will complete a short questionnaire to check the inclusion criterion, the results of the measurement of follicle count and hormone measurement (including AMH). Cases and controls will respond to self-administered questionnaire at inclusion with information about their medical history, their demographics, their tobacco and alcohol consumption, their occupation and products handled in the workplace. Blood samples (for measure of persistent organic pollutants and heavy metals) and urine (for measure of metabolites of glycol ethers) will be collect at baseline. Occupational exposures to solvents will be defined using job exposures matrices. The risk of decreased ovarian reserve will be analyzed using logistic regressions for each exposure of interest adjusting for potential confounders.
  Interventions: Other: Self-administered questionnaire and blood and urine samples

INTERVENTIONS:
Other: Self-administered questionnaire and blood and urine samples — Self-administered questionnaire and blood and urine samples

SUMMARY:
Early ovarian reserve decreased is one of the main causes of infertility for women after 35 years. The relationship between this decreased and exposure to chemicals, including persistent endocrine disruptors or organic solvents, has been little studied. However, several in vivo or in vitro experimental studies suggested that these chemicals may impaired ovarian function.

The main objective is to study the relationship between early ovarian reserve decreased and exposure to persistent organic pollutants.

The secondary objectives are to study the relationship between early ovarian reserve decreased and exposure to organic solvents and heavy metals.

Multicenter case-control study. This project will permit to increase the knowledge concerning the etiology of early decreased ovarian reserve. Considering that exposure of interest are frequent, the results may be important in a public health perspective. If associations are observed in this study, the results may encouraged prevention strategy.

DETAILED DESCRIPTION:
Cases and controls will benefit, as usual in France concerning infertility etiology examinations, of a follicle antral count by transvaginal ultrasound and AMH measurement.

At baseline, physicians will complete a short questionnaire to check the inclusion criterion, the results of the measurement of follicle count and hormone measurement (including AMH). Cases and controls will respond to self-administered questionnaire at inclusion with information about their medical history, their demographics, their tobacco and alcohol consumption, their occupation and products handled in the workplace. Blood samples (for measure of persistent organic pollutants and heavy metals) and urine (for measure of metabolites of glycol ethers) will be collect at baseline. Occupational exposures to solvents will be defined using job exposures matrices. The risk of decreased ovarian reserve will be analyzed using logistic regressions for each exposure of interest adjusting for potential confounders.

ELIGIBILITY:
Inclusion Criteria :

The cases will be:

* women among couples consulting for infertility in 4 centers for medically assisted procreation (AMP) performing in vitro fertilization in the Brittany Pays de Loire region: the university hospital (CHU) of BREST, the CHU of RENNES, the La Sagesse clinic in RENNES and the CHU de NANTES,
* having at least one characteristic of alteration of the ovarian reserve: a total number of antral follicles (left ovary + right ovary) less than 7 and / or a blood level of anti-Müllerian hormone (AMH) less than or equal to 1 , 1 ng / ml,
* age between 18 and 40 years old,
* with, in the event of past stimulation, at least one month since the last stimulation at the time of the blood and urine samples,
* having signed a free and informed consent.

For each case, two controls will be included with a pairing on the center and on the age group of 5 years (frequency pairing). It will be :

* women among couples consulting for infertility in 4 centers for medically assisted procreation (AMP) performing in vitro fertilization in the Brittany Pays de Loire region: the university hospital (CHU) of BREST, the CHU of RENNES, the La Sagesse clinic in RENNES and the CHU de NANTES,
* whose infertility assessment is strictly normal (AMH between 1.5 and 5 ng / ml, without genital malformation and with a menstrual cycle between 26 and 35 days),
* age between 18 and 40 years old,
* with, in the event of past stimulation, at least one month since the last stimulation at the time of the blood and urine samples,
* having signed a free and informed consent.

The non-inclusion criteria for cases and witnesses will be:

* ovarian endometriosis,
* polycystic ovary syndrome,
* a history of adnexal surgery,
* a history of cancer with chemotherapy or radiotherapy,
* morbid obesity (BMI ≥ 35 kg / m²),
* a chromosomal genetic syndrome (Turner and Fragile X)
* adults who are the subject of legal protection (safeguard of justice, curatorship, guardianship) and persons deprived of their liberty.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 335 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Persistant organic pollutants dosage | Day 1
  Persistant organic pollutants levels

SECONDARY OUTCOMES:
Organic solvents dosage | Day 1
  Occupational exposure to organic solvents
Glycol ethers métabolites dosage | Day 1
  Occupational exposure to glycol ethers metabolites.
Heavy metals dosage | Day 1
  Occupational exposure to heavy metals.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Brest university hospital, Brest
  - Nantes university hospital, Nantes
  - Cabinet de Gynécologie Malakoff, Rennes
  - Clinique Mutualiste de La Sagesse, Rennes
  - Rennes university hospital, Rennes

REFERENCES:
- [Result] Genard-Walton M, Warembourg C, Duros S, Mercier F, Lefebvre T, Guivarc'h-Leveque A, Le Martelot MT, Le Bot B, Jacquemin B, Chevrier C, Cordier S, Costet N, Multigner L, Garlantezec R. Serum persistent organic pollutants and diminished ovarian reserve: a single-exposure and mixture exposure approach from a French case-control study. Hum Reprod. 2023 Apr 3;38(4):701-715. doi: 10.1093/humrep/dead028. PMID 36881900